CLINICAL TRIAL: NCT03822195
Title: Evaluation of Lectine Pathway in Assessment of Unstable Carotid Plaque
Brief Title: Lectine Pathway in Unstable Carotid Plaque
Status: Withdrawn | Type: Observational
Why Stopped: PI changed Institution
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Angela M.R. Ferrante, Angela M.R. Ferrante MD PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2124
Record Dates: First submitted 2019-01-07; First posted 2019-01-30 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Carotid Artery Plaque; Mannose-Binding Lectin Complement Pathway
Keywords: carotid artery atherosclerosis; alternative complement pathway
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Atherosclerotic plaque surgically removed from the carotid bifurcation Peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- asymptomatic: asymptomatic patients undergoing carotid endoarterectomy for stenosis >70% (velocimetric criteria at echodoppler)
  Interventions: Procedure: Carotid endoarterectomy
- symptomatic: symptomatic (TIA, crescendo TIA, minor stroke) patients undergoing carotid endoarterectomy, independently from stenosis evaluated by echodoppler
  Interventions: Procedure: Carotid endoarterectomy

INTERVENTIONS:
Procedure: Carotid endoarterectomy — Surgical removal of carotid bifurcation plaque and arterial repair (direct suture or patch)
  Other Names: CEA

SUMMARY:
The study is aimed to investigate the possible role of lectin pathway - an alternative pathway of complement activation - in affecting stability of carotid atherosclerotic plaques and the possible correlations with clinical neurologic features.

DETAILED DESCRIPTION:
In addition to the known hemodynamic criteria, instable carotid plaques can be responsible for brain ischemia, therefore is paramount to identify preoperatively possible markers of plaque instability. The study is aimed to investigate the possible role of lectin pathway - an alternative pathway of complement activation - in affecting stability of carotid atherosclerotic plaques and the possible correlations with clinical neurologic features. Study population will include 40 patients with internal carotid artery stenosis >=70% (assessed by echocolordoppler), symptomatic or asymptomatic, surgically treated by endoarterectomy. Removed plaques will be evaluated by histologic exam and immunofluorescence for ficolins 1-2-3 and Mannose Binding Lectin (MBL). Plasma samples will be used for ELISA test of lectin pathway complement activation.

ELIGIBILITY:
Inclusion Criteria:

* patients undergone elective or urgent carotid endoarterectomy (CEA) for internal carotid stenosis >70% (assessed by velocimetric criteria) with or without neurologic symptoms

Exclusion Criteria:

* recent (<20 days) major/minor stroke with positive CT scan
* absolute contraindications to surgery (cardiac, respiratory, anesthesiologic risk)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include 40 patients with symptomatic or asymptomatic internal carotid artery stenosis >=70% (measured by echocolordoppler) treated by elective or urgent endoarterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
lectine pathway of complement activation in carotid plaques | preoperative
  assessment of association between plasmatic levels of complement activators and plaque instability (histologic index). Protein plasma levels will be assessed as optical density. Plaque instability will be quantified by a vulnerability score that combines four different histological parameters according to their quartile distribution (Fumagalli et al., Frontiers Immunology 2017). Their association will be analyzed as odds ratio (95%-CI) by a Fisher test.

SECONDARY OUTCOMES:
focal neurologic symptoms and plasmatic levels of complement activators | preoperative, postoperative day 3, 3 months after surgery
  Correlation of onset of focal neurologic symptoms (TIA, any stroke) due to carotid stenosis and peripheral plasma levels of complement activators. Neurological exam + CT or MNR will be used as clinical measurement tool
focal neurologic symptoms and histologic index of plaque instability | through study completion (average 1 year)
  correlation of onset of focal neurologic symptoms (TIA, any stroke) due to carotid stenosis and histologic index for plaque instability. Protein plasma levels will be assessed as optical density. Plaque instability will be quantified by a vulnerability score that combines four different histological parameters according to their quartile distribution (Fumagalli et al., Frontiers Immunology 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Angela MR Ferrante, MD, Principal Investigator — Fondazione Policlinico Universitario A.Gemelli IRCCS Roma

REFERENCES:
- [Background] Verhoeven B, Hellings WE, Moll FL, de Vries JP, de Kleijn DP, de Bruin P, Busser E, Schoneveld AH, Pasterkamp G. Carotid atherosclerotic plaques in patients with transient ischemic attacks and stroke have unstable characteristics compared with plaques in asymptomatic and amaurosis fugax patients. J Vasc Surg. 2005 Dec;42(6):1075-81. doi: 10.1016/j.jvs.2005.08.009. PMID 16376194
- [Background] Longhi L, Orsini F, De Blasio D, Fumagalli S, Ortolano F, Locatelli M, Stocchetti N, De Simoni MG. Mannose-binding lectin is expressed after clinical and experimental traumatic brain injury and its deletion is protective. Crit Care Med. 2014 Aug;42(8):1910-8. doi: 10.1097/CCM.0000000000000399. PMID 24810526
- [Background] Fust G, Munthe-Fog L, Illes Z, Szeplaki G, Molnar T, Pusch G, Hirschberg K, Szegedi R, Szeplaki Z, Prohaszka Z, Skjoedt MO, Garred P. Low ficolin-3 levels in early follow-up serum samples are associated with the severity and unfavorable outcome of acute ischemic stroke. J Neuroinflammation. 2011 Dec 29;8:185. doi: 10.1186/1742-2094-8-185. PMID 22206485
- [Background] Osthoff M, Katan M, Fluri F, Schuetz P, Bingisser R, Kappos L, Steck AJ, Engelter ST, Mueller B, Christ-Crain M, Trendelenburg M. Mannose-binding lectin deficiency is associated with smaller infarction size and favorable outcome in ischemic stroke patients. PLoS One. 2011;6(6):e21338. doi: 10.1371/journal.pone.0021338. Epub 2011 Jun 21. PMID 21712986
- [Background] Zangari R, Zanier ER, Torgano G, Bersano A, Beretta S, Beghi E, Casolla B, Checcarelli N, Lanfranconi S, Maino A, Mandelli C, Micieli G, Orzi F, Picetti E, Silvestrini M, Stocchetti N, Zecca B, Garred P, De Simoni MG; LEPAS group. Early ficolin-1 is a sensitive prognostic marker for functional outcome in ischemic stroke. J Neuroinflammation. 2016 Jan 20;13:16. doi: 10.1186/s12974-016-0481-2. PMID 26792363
- [Background] Pilely K, Fumagalli S, Rosbjerg A, Genster N, Skjoedt MO, Perego C, Ferrante AMR, De Simoni MG, Garred P. C-Reactive Protein Binds to Cholesterol Crystals and Co-Localizes with the Terminal Complement Complex in Human Atherosclerotic Plaques. Front Immunol. 2017 Aug 29;8:1040. doi: 10.3389/fimmu.2017.01040. eCollection 2017. PMID 28900428
- [Background] Hellings WE, Pasterkamp G, Vollebregt A, Seldenrijk CA, De Vries JP, Velema E, De Kleijn DP, Moll FL. Intraobserver and interobserver variability and spatial differences in histologic examination of carotid endarterectomy specimens. J Vasc Surg. 2007 Dec;46(6):1147-54. doi: 10.1016/j.jvs.2007.08.018. Epub 2007 Oct 22. PMID 17950565
- [Result] Fumagalli S, Perego C, Zangari R, De Blasio D, Oggioni M, De Nigris F, Snider F, Garred P, Ferrante AM, De Simoni MG. Lectin Pathway of Complement Activation Is Associated with Vulnerability of Atherosclerotic Plaques. Front Immunol. 2017 Mar 16;8:288. doi: 10.3389/fimmu.2017.00288. eCollection 2017. PMID 28360913